CLINICAL TRIAL: NCT05332054
Title: An Observational Long-Term Follow-up Study of Patients Who Received Prior Caribou Cell Therapy
Brief Title: Long-Term Follow-up Study
Acronym: LTFS
Status: Enrolling by invitation | Type: Observational
Sponsor: Caribou Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: LTFS
Record Dates: First submitted 2022-03-21; First posted 2022-04-18 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Lymphoma, Non-Hodgkin; Relapsed Non-Hodgkin Lymphoma; Refractory B-Cell Non-Hodgkin Lymphoma; Non-Hodgkin Lymphoma; Lymphoma; B Cell Lymphoma; B-Cell Non-Hodgkin's Lymphoma; Hematologic Malignancy; Relapsed/Refractory Multiple Myeloma; Relapsed/Refractory Acute Myeloid Leukemia
Keywords: Allogeneic CAR-T; CB-010; CB-011; CB-012
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, B-Cell; Lymphoma; Hematologic Neoplasms; Multiple Myeloma; Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who received IP in a Caribou-sponsored, special access program or IIT and provided informed: consent for the LTFS
  Interventions: Biological: Caribou-sponsored investigational therapy

INTERVENTIONS:
Biological: Caribou-sponsored investigational therapy — N/A this is an observational study

SUMMARY:
This is an observational, non-interventional, LTFS of investigational Caribou therapies in patients who have participated in a parent study: a prior Caribou-sponsored clinical study, special access program, or an IIT. The objective is to evaluate the long-term safety, through 15 years post infusion, in patients who received IPs in a Caribou-sponsored clinical study, special access program or IIT.

DETAILED DESCRIPTION:
This is an observational, non-interventional, LTFS of investigational Caribou therapies in patients who have participated in a parent study: a prior Caribou-sponsored clinical study, special access program, or an IIT. The objective is to evaluate the long-term safety, through 15 years post infusion, in patients who received IPs in a Caribou-sponsored clinical study, special access program or IIT.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent (by patient or legal representative) obtained prior to study-specific activities/enrollment
* Completed a Caribou-sponsored study or was administered Caribou IP under a special access program or as part of an IIT
* Use of an effective method of birth control by women of childbearing potential and their partners and men with partners of childbearing potential (partners must also use an effective birth control method) through 12 months post IP infusion.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who received IP in a Caribou-sponsored clinical study, special access program, or IIT and provided informed consent for the LTFS
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-03-16 (Actual); Primary Completion 2041-12 (Estimated); Study Completion 2041-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of targeted NSAEs | 15 Years
  Incidence of targeted NSAEs
Frequency of targeted NSAEs | 15 Years
  Frequency of targeted NSAEs
Duration of targeted NSAEs | 15 Years
  Duration of targeted NSAEs
Outcome of targeted NSAEs | 15 Years
  Outcome of targeted NSAEs
Incidence of AESIs | 15 Years
  Incidence of AESIs
Frequency of AESIs | 15 Years
  Frequency of AESIs
Duration of AESIs | 15 Years
  Duration of AESIs
Outcome of AESIs | 15 Years
  Outcome of AESIs
Incidence of targeted SAEs | 15 Years
  Incidence of targeted SAEs
Frequency of targeted SAEs | 15 Years
  Frequency of targeted SAEs
Duration of targeted SAEs | 15 Years
  Duration of targeted SAEs
Outcome of targeted SAEs | 15 Years
  Outcome of targeted SAEs
Incidence of AEs related to IP leading to death | 15 Years
  Incidence of AEs related to IP leading to death

SECONDARY OUTCOMES:
Overall survival | 15 years
  Assessment of overall survival and disease progression as described in the SOA

CONTACTS AND LOCATIONS:
Locations (30):
- United States (30):
  - University of Alabama, Birmingham, Alabama
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Honor Health Research Institute, Scottsdale, Arizona
  - University of California Irvine, Irvine, California
  - University of California San Diego, La Jolla, California
  - University of Colorado, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - University of Miami, Miami, Florida
  - AdventHealth Medical Group Blood & Marrow Transplant at Orlando, Orlando, Florida
  - Blood & Marrow Transplant Group of Georgia, Atlanta, Georgia
  - Augusta University/Georgia Cancer Center, Augusta, Georgia
  - University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - University of Kentucky, Lexington, Kentucky
  - Norton Cancer Institute, Louisville, Kentucky
  - Regional Cancer Care Associates - Hackensack, Hackensack, New Jersey
  - Atlantic Health System Cancer Care, Morristown, New Jersey
  - Weill Cornell Medicine, New York, New York
  - Icahn School of Medicine at Mt. Sinai, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Levine Cancer Center, Charlotte, North Carolina
  - Oncology Hematology Care, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute - TriStar Health, Nashville, Tennessee
  - Baylor Research Institute, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute at the University of Utah, Salt Lake City, Utah
  - Virginia Commonwealth University, Richmond, Virginia
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided